CLINICAL TRIAL: NCT01626846
Title: Cognitive Impairments, Self-Esteem & Academic Performance in Teenagers With Neurofibromatosis Type 1
Brief Title: How Neurofibromatosis Type 1 (NF1) Affects Schoolwork and Self-Esteem
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: John Jay High School (Other)
Responsible Party: Sponsor
Other Study IDs: NF Survey 2012
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NF1 teenagers

SUMMARY:
The study will seek to determine whether there is a corresponding deficit in school performance for teenagers with NF1. Secondly, the study seeks to explore the issue of self-esteem in teenagers with NF1.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Neurofibromatosis Type 1

Exclusion Criteria:

* Neurofibromatosis Type 2
* Schwannomatosis

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Teenagers aged 14-17 years with NF1
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Evidence of effect on self-esteem evidenced by self-esteem scores | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Karlik, PhD, Study Director — Westchester Community College
Locations (1):
- John Jay High School, Cross River, New York, United States